CLINICAL TRIAL: NCT02135445
Title: A Phase 2, Randomized, Open-Label, Parallel Group Study Evaluating the Safety and Efficacy of TAK-385, an Oral Gonadotropin-Releasing Hormone (GnRH) Antagonist, for Patients With Localized Prostate Cancer Requiring Neoadjuvant and Adjuvant Androgen Deprivation Therapy With External Beam Radiation Therapy (EBRT)
Brief Title: Safety and Efficacy of TAK-385 for Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C27003 Merge to Takeda; U1111-1152-9537 (Other: World Health Organization); 2013-005002-53 (EudraCT Number); 14/LO/1052 (Registry Identifier: NRES)
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer
Keywords: Drug therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — relugolix; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAK-385 (Experimental): TAK-385 320 mg, tablets, orally, once, on Day 1, followed by TAK-385 120 mg, orally, once daily for 24 weeks. Each participant may have one upward dose adjustment of 40 mg for efficacy and/or one downward dose adjustment of 40 mg for safety during the study.
  Interventions: Drug: TAK-385
- Degarelix (Active Comparator): Degarelix 240 mg, injection, subcutaneous, on Day 1, followed by degarelix 80 mg, injection, subcutaneous, once every four weeks, for 24 weeks.
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: TAK-385 — TAK-385 tablet
  Arms: TAK-385
Drug: Degarelix — Degarelix injection
  Other Names: Firmagon®
  Arms: Degarelix

SUMMARY:
The purpose of this study is to evaluate the efficacy of TAK-385 for achieving and maintaining testosterone suppression.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-385. Men with prostate cancer benefit from receiving androgen deprivation therapy (ADT) to minimize testosterone levels before, during and after EBRT. This combination increases the potential success of treating their disease. This study will see if TAK-385 [an oral gonadotropin-releasing hormone (GnRH) antagonist] brings testosterone levels down sufficiently, with the convenience and comfort of taking a pill. It will look at the time it takes to restore testosterone levels after radiation therapy as well. One hundred participants will be assigned by chance (like flipping a coin) to a treatment group: 60 to TAK-385, and 40 to degarelix.

Those assigned to TAK-385 will take a daily pill. Those assigned to degarelix will receive an injection under the skin once every four weeks at the clinic. They will start radiation therapy when testosterone is low enough, after at least 12 weeks of treatment. This trial will be conducted at clinics in the United States (US) and United Kingdom (UK). Participants will visit the clinic up to 14 times over 37 weeks for physical exams and blood tests, and might receive one follow-up telephone call.

ELIGIBILITY:
Inclusion Criteria:

1. Is male, 18 years of age or older.
2. Has histologically confirmed diagnosis of localized prostate adenocarcinoma of intermediate risk for which 6-month neoadjuvant and adjuvant androgen deprivation therapy (ADT) to EBRT is indicated. Intermediate risk per National Comprehensive Cancer Network (NCCN) guidelines includes one of the following:

   1. T2b-T2c disease, or
   2. Gleason score 7, or
   3. Prostate-specific antigen (PSA) 10-20 nanogram per milliliter (ng/mL).
3. Is scheduled for EBRT to begin greater than or equal to (>=) 12 weeks after the Baseline visit.
4. Has serum testosterone at screening greater then (>) 150 nanogram per deciliter (ng/dL) (5.2 nanomoles per liter [nmol/L]).
5. Has screening serum PSA concentration >2 ng/mL.
6. Has body mass index (BMI) >=18.0 at screening or baseline.
7. Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at screening or baseline.
8. Is a male participant, even if surgically sterilized (that is, status postvasectomy), who: Agrees to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or, Agrees to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception.).
9. Has given voluntary written consent before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
10. Has suitable venous access for the study-required blood sampling, including pharmacokinetic (PK) and pharmacodynamic sampling.

Exclusion Criteria:

1. Has metastatic disease (based on investigator evaluation and assuming no likely metastatic pelvic lymph nodes >1.0 cm in long axis diameter).
2. Had prior or current use of a gonadotropin-releasing hormone (GnRH) analog or androgen receptor antagonist as first-line hormone therapy, unless total use was less than 6 months and not more recently than 1 year before the planned baseline visit.
3. Had diagnosis of or treatment for another malignancy within 2 years before the first dose of study drug, or previous diagnosis of another malignancy with evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
4. Has abnormal screening and/or baseline laboratory values that suggest a clinically significant underlying disease, or the following laboratory values:

   1. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 * institutional upper limit of the normal range (ULN);
   2. Serum creatinine >2.0 milligram per deciliter (mg/dL);
   3. Total bilirubin >2.0 * institutional ULN (unless documented Gilbert's disease);
   4. Uncontrolled diabetes (Hemoglobin A1c [HbA1c] >10 [percent] %) or previously undiagnosed diabetes mellitus with HbA1c >8%.
5. Has history of myocardial infarction, unstable symptomatic ischemic heart disease, any ongoing cardiac arrhythmias of Grade >2 (chronic stable atrial fibrillation on stable anticoagulant therapy is allowed), thromboembolic events (example, deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events), or any other significant cardiac condition (example, pericardial effusion, restrictive cardiomyopathy) within 6 months before receiving the first dose of study drug.
6. Has electrocardiogram (ECG) abnormalities of:

   1. Q-wave infarction, unless identified 6 or more months before screening;
   2. Heart rate-corrected QT interval millisecond (msec) (QTcF interval) >480 msec. If QTcF is prolonged in a participant with a pacemaker, the participant may be enrolled in the study upon discussion with the project clinician;
   3. If the QTcF interval is 450-480 msec, inclusive, in a participant with current use of medications with known effects on QT interval, the participant may be enrolled in the study following discussion with the project clinician.
7. Has congenital long QT syndrome.
8. Is currently using Class IA (example, quinidine, procainamide) or Class III (example, amiodarone, sotalol) antiarrhythmic medications.
9. Has uncontrolled hypertension despite appropriate medical therapy (sitting blood pressure [BP] of greater than 160 millimeters of mercury (mmHg) systolic and 90 mmHg diastolic at 2 separate measurements no more than 60 minutes apart during the Screening visit). Participants with systolic BP measurements >160 mmHg may be rescreened. Participants with systolic BP measurements 141-160 mmHg, although eligible, should be referred for further management of hypertension if indicated.
10. Has known, previously diagnosed human immunodeficiency virus (HIV) infection, active chronic hepatitis B or C, life-threatening illness unrelated to prostate cancer, or any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with participation in this study. Specific screening for chronic viral illness is at the discretion of the site and/or local institutional review board (IRB).
11. Has received treatment with any investigational products within 3 months before the first dose of study drug.
12. Is a primary family member (spouse, parent, child, or sibling) of anyone involved in the conduct of the study or is a study site employee.
13. Has known gastrointestinal (GI) disease, condition or procedure that could interfere with the oral absorption or tolerance of TAK-385, including difficulty swallowing tablets.
14. Is using any medication or food products listed in the excluded medications and dietary products table within 2 weeks before the first dose of study drug. This list includes moderate and strong inhibitors or inducers of cytochrome P450 (CYP3A4/5) and P-glycoprotein (P-gp). Participants must have no history of amiodarone use in the 6 months before the first dose of TAK-385.
15. Has admission or evidence of alcohol or drug abuse or use of illicit drugs.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (25):
- United States (19):
  - Birmingham, Alabama
  - San Diego, California
  - Denver, Colorado
  - Bradenton, Florida
  - Daytona Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Plantation, Florida
  - Jeffersonville, Indiana
  - Wichita, Kansas
  - Shreveport, Louisiana
  - Omaha, Nebraska
  - Syracuse, New York
  - Columbus, Ohio
  - Eugene, Oregon
  - Myrtle Beach, South Carolina
  - Dallas, Texas
  - San Antonio, Texas
  - Virginia Beach, Virginia
- United Kingdom (6):
  - Brighton, East Sussex
  - Manchester, Greater Manchester
  - Metropolitan Borough of Wirral, Merseyside
  - Taunton, Somerset
  - Sutton, Surrey
  - Birmingham, West Midlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 23 investigative sites in the United States (US) and the United Kingdom (UK).
Pre-assignment Details: Participants with a diagnosis of localized prostate cancer were enrolled in 1 of the 2 treatment groups to receive TAK-385 120 milligram (mg) or degarelix 80 mg.
Groups:
- Experimental: TAK-385 120 mg: TAK-385 320 mg, tablets, orally, as loading dose on Day 1 followed by TAK-385 120 mg, tablets, orally, daily as maintenance dose starting from Day 2 up to Day 7 Week 24.
- Experimental: Degarelix 80 mg: Degarelix 240 mg, injection, subcutaneously, on Day 1 Week 1 followed by Degarelix 80 mg, injection, subcutaneously, once every 4 weeks beginning on Day 1 Week 5 up to Day 1 Week 21.
Period: Overall Study
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Started | 65 | 38
Completed | 63 | 38
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg | Total
Number analyzed (Participants) | 65 | 38 | 103
Age, Customized [Number; unit: participants]
  18 to 64 years | 9 | 7 | 16
  65 to 84 years | 55 | 31 | 86
  Greater than or equal to (>=) 85 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 65 | 38 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 62 | 35 | 97
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 58 | 31 | 89
  Black or African American | 7 | 7 | 14
Eastern Cooperative Oncology Group (ECOG) Performance status [Number; unit: participants] — ECOG assessed participants performance status on a 6-point scale: 0: Fully active, able to carry on all predisease performance without restriction; 1: Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature; 2: Ambulatory, capable of selfcare, unable to carry out any work activities, up and about greater than (>)50 percent (%) of waking hours; 3:Capable of limited selfcare,confined to bed or chair >50% of waking hours; 4: Completely disabled, not capable of any selfcare, totally confined to bed or chair; 5:Dead.
  participants
    Grade 0 | 60 | 33 | 93
    Grade 1 | 4 | 4 | 8
    Missing | 1 | 1 | 2
Prostate Cancer Type [Number; unit: participants]
  Adenocarcinoma insitu,Not otherwise specified(NOS) | 5 | 1 | 6
  Adenocarcinoma, NOS | 59 | 37 | 96
  Other | 1 | 0 | 1
Primary Gleason Score [Number; unit: participants] — Gleason score is a histological score that, together with other clinical factors may be used to predict the potential aggressiveness of the cancer and thus its risk of eventually spreading. Gleason scores range from 2-10, where 2-4: lower risk; 5-6: moderate risk; 8-10: higher risk with lower score representing most well-differentiated tumors and higher score representing least-differentiated tumors. Primary grading in Gleason score is assigned to dominant pattern of tumor which has to be >50% of total pattern seen.
  participants
    Primary grade 3 | 28 | 18 | 46
    Primary grade 4 | 24 | 15 | 39
    Primary grade missing | 13 | 5 | 18
Secondary Gleason Score [Number; unit: participants] — Gleason score is a histological score that, together with other clinical factors may be used to predict the potential aggressiveness of the cancer and thus its risk of eventually spreading. Gleason scores range from 2-10, where 2-4: lower risk; 5-6: moderate risk; 8-10: higher risk with lower score representing most well-differentiated tumors and higher score representing least-differentiated tumors. Primary grading in Gleason score is assigned to dominant pattern of tumor which has to be >50% of total pattern seen.
  participants
    Secondary grade 3 | 22 | 12 | 34
    Secondary grade 4 | 28 | 19 | 47
    Secondary grade 5 | 2 | 2 | 4
    Secondary grade missing | 13 | 5 | 18
Total Gleason Score [Number; unit: participants] — Gleason score is a histological score that, together with other clinical factors may be used to predict the potential aggressiveness of the cancer and thus its risk of eventually spreading. Gleason scores range from 2-10, where 2-4: lower risk; 5-6: moderate risk; 8-10: higher risk with lower score representing most well-differentiated tumors and higher score representing least-differentiated tumors. Primary grading in Gleason score is assigned to dominant pattern of tumor which has to be >50% of total pattern seen.
  participants
    Total Gleason score 6 | 5 | 2 | 7
    Total Gleason score 7 | 40 | 26 | 66
    Total Gleason score 8 | 5 | 3 | 8
    Total Gleason score 9 | 2 | 2 | 4
    Total Gleason score missing | 13 | 5 | 18
Initial diagnosis of Primary Tumor (T) [Number; unit: participants] — TNM Stages: T1: unapparent neither palpable nor visible by imaging, T1a: histologic finding in 5% or less of tissue resected, T1b: histological finding in >5% of tissue resected, T1c: identified by needle biopsy, T2: confined within prostate, T2a: one-half of one lobe or less, T2b: involves more than one-half of one lobe but not both lobes, T2c: involves both lobes, T3: extends through prostate capsule, T3a: Extracapsular extension Including microscopic bladder neck involvement, T3b: invades seminal vesicles, T4: fixed or invades adjacent structures other than seminal vesicles
  participants
    T1 | 2 | 3 | 5
    T1a | 0 | 1 | 1
    T1c | 24 | 16 | 40
    T2 | 4 | 4 | 8
    T2a | 13 | 2 | 15
    T2b | 7 | 2 | 9
    T2c | 8 | 7 | 15
    T3 | 0 | 2 | 2
    Not available | 7 | 1 | 8
Initial diagnosis: Regional Lymph Nodes (N) [Number; unit: participants] — TNM: Regional lymph nodes (N) staging included NX: Regional lymph nodes were not assessed, and N0: No regional lymph node metastasis.
  participants
    N0 | 41 | 18 | 59
    NX | 16 | 18 | 34
    Not available | 8 | 2 | 10
Initial diagnosis: Distant Metastasis (M) [Number; unit: participants] — TNM: Distant metastasis stages included, M0: No distant metastasis.
  participants
    M0 | 56 | 34 | 90
    Not available | 9 | 4 | 13
Diagnosis of Primary Tumor at Study entry [Number; unit: participants] — TNM Stages: T1: unapparent neither palpable nor visible by imaging, T1a: histologic finding in 5% or less of tissue resected, T1b: histological finding in >5% of tissue resected, T1c: identified by needle biopsy, T2: confined within prostate, T2a: one-half of one lobe or less, T2b: involves more than one-half of one lobe but not both lobes, T2c: involves both lobes, T3: extends through prostate capsule, T3a: Extracapsular extension Including microscopic bladder neck involvement, T3b: invades seminal vesicles, T4: fixed or invades adjacent structures other than seminal vesicles
  participants
    T1 | 1 | 1 | 2
    T1a | 0 | 1 | 1
    T1c | 20 | 10 | 30
    T2 | 6 | 5 | 11
    T2a | 12 | 3 | 15
    T2b | 7 | 1 | 8
    T2c | 7 | 7 | 14
    T3 | 0 | 1 | 1
    T3a | 1 | 0 | 1
    TX | 0 | 1 | 1
    Not available | 11 | 8 | 19
Study entry: N [Number; unit: participants] — TNM: Regional lymph nodes staging included NX: Regional lymph nodes were not assessed, and N0: No regional lymph node metastasis.
  participants
    N0 | 39 | 19 | 58
    NX | 13 | 10 | 23
    Not available | 13 | 9 | 22
Study entry: M [Number; unit: participants] — TNM: Distant metastasis stages included, M0: No distant metastasis.
  participants
    M0 | 51 | 28 | 79
    Not available | 14 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Effective Castration Rate Over 25 Weeks
Description: Castration rate is defined as the observed percentage of participants who have testosterone concentrations less than (<) 50 nanogram per deciliter (ng/dL) (1.73 nanomole per liter [nmol/L]) at all scheduled visits.
Time Frame: Day 1 Week 5 up to Day 1 Week 25
Population: Safety population included all participants who received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
percentage of participants | 95 [87.1 to 99.0] | 89 [75.2 to 97.1]

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Vital Signs
Time Frame: Baseline up to Week 29
Population: Safety population included all participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
participants | 2 | 1

3. Secondary Outcome: Number of Participants With TEAEs Related to Physical Findings
Time Frame: Baseline up to Week 29
Population: Safety population included all participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
participants | 5 | 1

4. Secondary Outcome: Number of Participants With TEAEs Related to 12-lead Electrocardiogram (ECG) Findings
Time Frame: Baseline up to Week 29
Population: Safety population included all participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
participants | 1 | 1

5. Secondary Outcome: Number of Participants With TEAEs Categorized Into Investigations Related to Chemistry, Hematology or Urinalysis
Time Frame: Baseline up to Week 29
Population: Safety population included all participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
participants
  Liver function analyses | 0 | 6
  Reproductive hormone analyses | 2 | 4
  Carbohydrate tolerance analyses inclusive diabetes | 1 | 0
  Cell marker analyses | 0 | 1
  Platelet analyses | 0 | 1
  Red blood cell analyses | 1 | 0
  Skeletal and cardiac muscle analyses | 1 | 0
  Urinalysis not elsewhere classified (NEC) | 1 | 0

6. Secondary Outcome: Number of Participants Reporting One or More TEAEs and Serious Adverse Events (SAEs)
Time Frame: Baseline up to Week 29
Population: Safety population included all participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
participants
  TEAEs (including SAEs and non-SAEs) | 56 | 37
  SAEs | 1 | 3

7. Secondary Outcome: Average Percent Change in Prostate Size
Description: Percent change in prostate size was assessed at a follow up visit between Day 1 Week 9 to Day 1 Week 13.
Time Frame: Baseline, Day 1 Week 9 to Day 1 Week 13
Population: Safety population where baseline and post-baseline assessments were available. Safety population included all participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 57 | 38
percent change | -25.1 (20.03) | -27.2 (25.88)

8. Secondary Outcome: Time to Achieve Effective Castration
Description: Time to effective castration is defined as days from first dose to first testosterone measurement that is <50 ng/dL.
Time Frame: Baseline up to Week 37
Population: Safety population included all participants who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
days | 4 [2 to 4] | 3 [2 to 4]

9. Secondary Outcome: Time to Achieve Profound Castration
Description: Time to profound castration is defined as days from first dose to first testosterone measurement that is <20 ng/dL.
Time Frame: Baseline up to Week 37
Population: Safety population included all participants who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
days | 15 [8 to 15] | 12 [8 to 15]

10. Secondary Outcome: Estimated Time to Testosterone Recovery (TTR)
Description: TTR is defined as the time from 1 day after the last dose of TAK-385 or 4 weeks plus 1 day after the last dose of degarelix to testosterone recovery. Testosterone recovery is defined as back to baseline or >280 ng/dL whichever occurs first. TTR was determined during 12 weeks after the discontinuation of androgen deprivation therapy (ADT).
Time Frame: Up to Day 1 Week 37
Population: Safety population included all participants who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 6
days | 91 [62 to 127] | 100 [100 to 106]

11. Secondary Outcome: Percentage of Participants Who Have Recovered to Baseline Value of Testosterone
Time Frame: Up to Day 1 Week 37
Population: Safety population included all participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
percentage of participants | 25 | 11

12. Secondary Outcome: Percentage of Participants Who Have Recovered to >280 ng/dL Testosterone
Time Frame: Day 1 Week 25 up to Day 1 Week 37
Population: Safety population included all participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
percentage of participants | 48 | 13

13. Secondary Outcome: Number of Participants With PSA Response of >=50% and >=90% Reduction
Description: Prostate-specific Antigen (PSA) response was defined as 50% and 90% reduction from baseline in serum PSA levels.
Time Frame: Day 1 Week 13
Population: Safety population included all participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
participants
  >=50% reduction | 64 | 37
  >=90% reduction | 36 | 18

14. Secondary Outcome: Percent Change From Baseline in Serum PSA Concentration
Time Frame: Baseline, Day 1 of Week 2, 3 , 5, 9, 13, 17, 21, 25, 29, 33 and 37
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
percent change
  Day 1 Week 2: number analyzed (Participants) | 64 | 37
  Day 1 Week 2 | -29.348 (21.9312) | -26.756 (36.9407)
  Day 1 Week 3: number analyzed (Participants) | 65 | 37
  Day 1 Week 3 | -35.798 (48.5347) | -14.292 (108.1051)
  Day 1 Week 5: number analyzed (Participants) | 65 | 37
  Day 1 Week 5 | -60.519 (34.9460) | -64.509 (32.5843)
  Day 1 Week 9: number analyzed (Participants) | 62 | 37
  Day 1 Week 9 | -84.345 (13.7231) | -78.364 (42.6674)
  Day 1 Week 13: number analyzed (Participants) | 64 | 38
  Day 1 Week 13 | -88.065 (10.6750) | -85.735 (14.9181)
  Day 1 Week 17: number analyzed (Participants) | 64 | 37
  Day 1 Week 17 | -90.433 (10.0884) | -87.712 (13.8226)
  Day 1 Week 21: number analyzed (Participants) | 63 | 37
  Day 1 Week 21 | -95.837 (5.0062) | -94.347 (9.4243)
  Day 1 Week 25: number analyzed (Participants) | 64 | 37
  Day 1 Week 25 | -97.430 (3.3650) | -96.268 (7.6796)
  Day 1 Week 29: number analyzed (Participants) | 61 | 38
  Day 1 Week 29 | -96.614 (4.7552) | -96.858 (7.5198)
  Day 1 Week 33: number analyzed (Participants) | 62 | 38
  Day 1 Week 33 | -94.697 (6.4998) | -97.309 (7.3210)
  Day 1 Week 37: number analyzed (Participants) | 61 | 38
  Day 1 Week 37 | -94.998 (5.6555) | -97.144 (6.6127)

15. Secondary Outcome: PSA Nadir
Time Frame: Baseline up to Day 1 Week 25
Population: Safety population included all participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
microgram per liter (mcg/L) | 0.3 (0.72) | 0.3 (0.41)

16. Secondary Outcome: Serum PSA Concentration
Time Frame: Day 1 of Week 13, 25, 29, 33 and 37
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
mcg/L
  Day 1 Week 13: number analyzed (Participants) | 64 | 38
  Day 1 Week 13 | 1.104 (1.3287) | 1.486 (2.1381)
  Day 1 Week 25: number analyzed (Participants) | 64 | 37
  Day 1 Week 25 | 0.223 (0.3343) | 0.274 (0.4448)
  Day 1 Week 29: number analyzed (Participants) | 61 | 38
  Day 1 Week 29 | 0.268 (0.3357) | 0.211 (0.3653)
  Day 1 Week 33: number analyzed (Participants) | 62 | 38
  Day 1 Week 33 | 0.431 (0.5455) | 0.183 (0.3503)
  Day 1 Week 37: number analyzed (Participants) | 61 | 38
  Day 1 Week 37 | 0.410 (0.4635) | 0.210 (0.3325)

17. Secondary Outcome: Plasma Concentrations of TAK-385
Time Frame: Day 1 Week 1, 2, 3, 5, 9, 13, 17, 25, 33, 37: Pre-dose; Day 1 Week 5, 13: 2 hrs Post-dose; Day 4 Week 1: Pre-dose
Population: Safety population where TAK-385 assessments were available. Safety population included all participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Experimental: TAK-385 120 mg
Number analyzed (Participants) | 65
nanogram per milliliter (ng/mL)
  Day 1 Week 1: Predose | 0.1 (0.84)
  Day 1 Week 2: Predose: number analyzed (Participants) | 64
  Day 1 Week 2: Predose | 11.9 (19.69)
  Day 1 Week 3: Predose: number analyzed (Participants) | 64
  Day 1 Week 3: Predose | 10.4 (10.16)
  Day 1 Week 5: Predose | 9.3 (12.52)
  Day 1 Week 5: 2 hrs post-dose: number analyzed (Participants) | 62
  Day 1 Week 5: 2 hrs post-dose | 36.4 (38.14)
  Day 1 Week 9: Predose: number analyzed (Participants) | 63
  Day 1 Week 9: Predose | 11.4 (18.48)
  Day 1 Week 13: Predose: number analyzed (Participants) | 61
  Day 1 Week 13: Predose | 8.2 (6.25)
  Day 1 Week 13: 2 hrs post-dose: number analyzed (Participants) | 61
  Day 1 Week 13: 2 hrs post-dose | 35.8 (37.33)
  Day 1 Week 17: Predose: number analyzed (Participants) | 61
  Day 1 Week 17: Predose | 8.7 (7.44)
  Day 1 Week 25: Predose: number analyzed (Participants) | 60
  Day 1 Week 25: Predose | 9.5 (7.78)
  Day 1 Week 29: Predose: number analyzed (Participants) | 60
  Day 1 Week 29: Predose | 0.3 (0.38)
  Day 1 Week 33: Predose: number analyzed (Participants) | 62
  Day 1 Week 33: Predose | 0.1 (0.10)
  Day 1 Week 37: Predose: number analyzed (Participants) | 59
  Day 1 Week 37: Predose | 0.1 (0.05)
  Day 4 Week 1: Predose: number analyzed (Participants) | 59
  Day 4 Week 1: Predose | 10.5 (16.35)

18. Secondary Outcome: Serum Luteinizing Hormone (LH) Level
Time Frame: Baseline, Day 1 of Weeks 2, 3, 5, 9, 13, 17, 21, 25, 29, and 37
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milli-international units per milliliter
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
milli-international units per milliliter
  Baseline | 5.838 (5.0647) | 6.943 (7.6683)
  Day 1 Week 2: number analyzed (Participants) | 64 | 37
  Day 1 Week 2 | 0.388 (0.4167) | 0.539 (0.7122)
  Day 1 Week 3: number analyzed (Participants) | 65 | 37
  Day 1 Week 3 | 0.223 (0.3820) | 0.362 (0.5648)
  Day 1 Week 5: number analyzed (Participants) | 64 | 37
  Day 1 Week 5 | 0.178 (0.2547) | 0.252 (0.3280)
  Day 1 Week 9: number analyzed (Participants) | 64 | 36
  Day 1 Week 9 | 0.198 (0.4677) | 0.333 (0.5649)
  Day 1 Week 13: number analyzed (Participants) | 64 | 38
  Day 1 Week 13 | 0.180 (0.3979) | 0.265 (0.5073)
  Day 1 Week 17: number analyzed (Participants) | 64 | 37
  Day 1 Week 17 | 0.184 (0.3690) | 0.283 (0.5461)
  Day 1 Week 21: number analyzed (Participants) | 63 | 37
  Day 1 Week 21 | 0.199 (0.4670) | 0.294 (0.5523)
  Day 1 Week 25: number analyzed (Participants) | 64 | 37
  Day 1 Week 25 | 0.325 (0.7243) | 0.342 (0.6248)
  Day 1 Week 29: number analyzed (Participants) | 61 | 38
  Day 1 Week 29 | 4.204 (3.3259) | 0.464 (0.5756)
  Day 1 Week 37: number analyzed (Participants) | 62 | 38
  Day 1 Week 37 | 9.441 (5.6144) | 1.036 (1.4907)

19. Secondary Outcome: Serum Follicle-Stimulating Hormone (FSH) Level
Time Frame: Baseline, Day 1 of Week 2, 5, 13, 25 and 29
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
International units per liter (IU/L)
  Baseline | 11.826 (17.3909) | 11.716 (14.7839)
  Day 1 Week 2: number analyzed (Participants) | 64 | 37
  Day 1 Week 2 | 2.363 (2.9647) | 2.519 (2.8180)
  Day 1 Week 5: number analyzed (Participants) | 64 | 37
  Day 1 Week 5 | 0.706 (0.9289) | 0.973 (1.0951)
  Day 1 Week 13: number analyzed (Participants) | 63 | 38
  Day 1 Week 13 | 0.849 (1.1728) | 1.108 (1.3469)
  Day 1 Week 25: number analyzed (Participants) | 64 | 38
  Day 1 Week 25 | 1.475 (2.1842) | 1.471 (1.7437)
  Day 1 Week 29: number analyzed (Participants) | 62 | 38
  Day 1 Week 29 | 7.427 (5.4105) | 2.032 (1.9114)

20. Secondary Outcome: Serum Sex Hormone-Binding Globulin (SHBG) Level
Time Frame: Baseline, Day 1 of Week 2, 5, 13, 25 and 29
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
nmol/L
  Baseline | 45.528 (21.3167) | 41.784 (17.8412)
  Day 1 Week 2: number analyzed (Participants) | 65 | 37
  Day 1 Week 2 | 49.474 (22.3975) | 43.386 (15.9911)
  Day 1 Week 5: number analyzed (Participants) | 65 | 37
  Day 1 Week 5 | 46.797 (22.6572) | 41.778 (15.7575)
  Day 1 Week 13: number analyzed (Participants) | 64 | 38
  Day 1 Week 13 | 46.083 (24.6853) | 42.992 (19.2416)
  Day 1 Week 25: number analyzed (Participants) | 64 | 37
  Day 1 Week 25 | 46.258 (25.0679) | 44.305 (22.2005)
  Day 1 Week 29: number analyzed (Participants) | 61 | 38
  Day 1 Week 29 | 43.329 (20.8000) | 42.739 (21.9110)

21. Secondary Outcome: Percent Change From Baseline in Aging Male's Symptoms (AMS) Total Scale Score
Description: AMS scale is a self-administered questionnaire used to 1) assess symptoms of aging (independent from those that are disease related) between groups of males under different conditions; 2) evaluate the severity of symptoms over time; and 3) measure changes before and after androgen therapy. Each question was answered between none (1) to extremely severe (5) for 17 items from psychological (5 items), somatic (7 items), and sexual (5 items) categories. Total score is sum of all the item scores and range from 17 (minimum) to 85 (maximum), where high score indicated high level of symptoms.
Time Frame: Day 1 of Weeks 5, 13, 25, 29, 33 and 37
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
percent change
  Day 1 Week 5: number analyzed (Participants) | 62 | 38
  Day 1 Week 5 | 17.347 (36.1328) | 19.194 (27.8573)
  Day 1 Week 13: number analyzed (Participants) | 61 | 37
  Day 1 Week 13 | 31.461 (41.4029) | 36.117 (33.8115)
  Day 1 Week 25: number analyzed (Participants) | 62 | 38
  Day 1 Week 25 | 43.558 (52.4934) | 48.158 (41.2365)
  Day 1 Week 29: number analyzed (Participants) | 62 | 38
  Day 1 Week 29 | 33.692 (44.8331) | 36.950 (34.4352)
  Day 1, Week 33: number analyzed (Participants) | 62 | 38
  Day 1, Week 33 | 24.273 (40.0869) | 40.227 (37.9232)
  Day 1 Week 37: number analyzed (Participants) | 62 | 38
  Day 1 Week 37 | 14.562 (30.0487) | 40.535 (35.3799)

22. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30) Score
Description: EORTC QLQ-C30 included 30 questions comprising 9 multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, nausea/vomiting), single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties) and a global health and QOL scale. Most questions used 4 point scale (1 'Not at all' to 4 'Very much'); 2 questions used 7-point scale (1 'Very poor' to 7 'Excellent'). All domain scores were calculated as an average of item scores and transformed to 0-100 score range where a high score from 0-100 indicates: A high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status/quality of life (QoL) represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problem.
Time Frame: Baseline and last post-baseline value up to Week 37
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
units on scale
  Day 1 Week 5: number analyzed (Participants) | 62 | 37
  Day 1 Week 5 | -5.10 (1.833) | -0.26 (2.370)
  Day 1 Week 13: number analyzed (Participants) | 61 | 37
  Day 1 Week 13 | -4.29 (1.837) | -4.33 (2.364)
  Day 1 Week 25: number analyzed (Participants) | 60 | 38
  Day 1 Week 25 | -10.04 (1.842) | -7.27 (2.349)
  Day 1 Week 29: number analyzed (Participants) | 62 | 38
  Day 1 Week 29 | -7.11 (1.826) | -8.14 (2.349)
  Day 1 Week 33: number analyzed (Participants) | 62 | 38
  Day 1 Week 33 | -6.24 (1.830) | -6.39 (2.349)
  Day 1 Week 37: number analyzed (Participants) | 62 | 38
  Day 1 Week 37 | -7.84 (1.833) | -6.61 (2.349)

23. Secondary Outcome: Change From Baseline in 25-item Prostate Cancer-specific Questionnaire Supplement (EORTC QLQ-PR25) Score
Description: EORTC QLQ-PR25 : EORTC module designed to supplement the QLQ-C30 for any application in prostate cancer. It Consist of 25 questions distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Questions used 4 point scale (1 'Not at all' to 4 'Very much'). All raw domain scores are linearly transformed to a 0-100 scale, with higher scores reflecting either more symptoms (urinary, bowel, hormonal treatment-related symptoms) or higher levels of activity or functioning (sexual).
Time Frame: Baseline and last post-baseline value up to Week 37
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Number analyzed (Participants) | 65 | 38
units on scale
  Sexual activity: Day 1 Week 5: number analyzed (Participants) | 62 | 37
  Sexual activity: Day 1 Week 5 | -9.78 (2.957) | -9.53 (3.823)
  Sexual activity: Day 1 Week 13: number analyzed (Participants) | 61 | 37
  Sexual activity: Day 1 Week 13 | -17.43 (2.967) | -11.54 (3.816)
  Sexual activity: Day 1 Week 25: number analyzed (Participants) | 60 | 38
  Sexual activity: Day 1 Week 25 | -19.32 (2.978) | -12.57 (3.784)
  Sexual activity: Day 1 Week 29: number analyzed (Participants) | 62 | 38
  Sexual activity: Day 1 Week 29 | -19.06 (2.948) | -5.12 (3.784)
  Sexual activity: Day 1 Week 33: number analyzed (Participants) | 62 | 38
  Sexual activity: Day 1 Week 33 | -12.40 (2.952) | -9.94 (3.784)
  Sexual activity: Day 1 Week 37: number analyzed (Participants) | 62 | 38
  Sexual activity: Day 1 Week 37 | -6.60 (2.957) | -6.00 (3.784)
  HTRS: Day 1 Week 5: number analyzed (Participants) | 62 | 37
  HTRS: Day 1 Week 5 | 6.55 (1.275) | 7.02 (1.651)
  HTRS: Day 1 Week 13: number analyzed (Participants) | 61 | 37
  HTRS: Day 1 Week 13 | 10.06 (1.275) | 9.98 (1.648)
  HTRS: Day 1 Week 25: number analyzed (Participants) | 60 | 38
  HTRS: Day 1 Week 25 | 13.34 (1.276) | 12.48 (1.641)
  HTRS: Day 1 Week 29: number analyzed (Participants) | 62 | 38
  HTRS: Day 1 Week 29 | 11.53 (1.270) | 10.43 (1.641)
  HTRS: Day 1 Week 33: number analyzed (Participants) | 62 | 38
  HTRS: Day 1 Week 33 | 9.62 (1.273) | 10.72 (1.641)
  HTRS: Day 1 Week 37: number analyzed (Participants) | 62 | 38
  HTRS: Day 1 Week 37 | 8.67 (1.276) | 11.31 (1.641)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of TAK-385 or 4 weeks plus 30 days after degarelix injection, whichever is applicable.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Experimental: TAK-385 120 mg | Experimental: Degarelix 80 mg
Serious Adverse Events (participants affected / at risk) | 1/65 | 3/38
Other Adverse Events (participants affected / at risk) | 56/65 | 37/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: TAK-385 120 mg (N=65) | Experimental: Degarelix 80 mg (N=38)
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: TAK-385 120 mg (N=65) | Experimental: Degarelix 80 mg (N=38)
Hot flush (Vascular disorders) | 37 | 23
Fatigue (General disorders) | 17 | 6
Cataract (Eye disorders) | 10 | 7
Diarrhoea (Gastrointestinal disorders) | 12 | 5
Nocturia (Renal and urinary disorders) | 9 | 5
Pollakiuria (Renal and urinary disorders) | 8 | 6
Dysuria (Renal and urinary disorders) | 5 | 6
Constipation (Gastrointestinal disorders) | 6 | 3
Dizziness (Nervous system disorders) | 6 | 2
Headache (Nervous system disorders) | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1
Blood testosterone increased (Investigations) | 2 | 4
Erectile dysfunction (Reproductive system and breast disorders) | 3 | 3
Micturition urgency (Renal and urinary disorders) | 5 | 1
Nasopharyngitis (Infections and infestations) | 4 | 2
Sinusitis (Infections and infestations) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.